CLINICAL TRIAL: NCT05180916
Title: Priming the Epileptic Brain - Determining the Effect of Temporarily Addition of Transcutaneous Vagal Nerve Stimulation When Starting an add-on AED (in This Case Brivaracetam) in Patients With Refractory Focal Epilepsy
Brief Title: Priming the Epileptic Brain: tVNS to Improve Efficacy of add-on AED in Patients With Focal Epilepsy
Acronym: PREP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eindhoven University of Technology (Other)
Collaborators: Clinical Trial Center Maastricht B.V. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PREP_001
Record Dates: First submitted 2021-07-02; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Focal Epilepsy
Keywords: vagus nerve stimulation
MeSH Terms: conditions — Epilepsies, Partial

STUDY DESIGN:
Intervention Model Description: Randomized Controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brivaracetam + Transcutaneous vagal nerve stimulation (Active Comparator): Start of Brivaracetam (treatment as usual), combined with tVNS in the first 3 months of treatment
  Interventions: Device: TVNS
- Brivaracetam (No Intervention): Start of Brivaracetam (treatment as usual)

INTERVENTIONS:
Device: TVNS — Cerbomed NEMOS
  Arms: Brivaracetam + Transcutaneous vagal nerve stimulation

SUMMARY:
The most prevalent neurological disorder with also immense burden of disease, epilepsy, is in over 30 percent of patients difficult to treat. The ideal treatment regime would give complete control of disease in an early stage, not only for patient well-being, but also to prevent the onset of persistent pathologic epileptic networks in the brain. The first step in treatment is the trial, and error, of multiple anti-epileptic drugs (AEDs), while invasive brain stimulation (BS) techniques with network modulating properties are saved as a last resort. The investigators hypothesize that pharmacotherapeutic treatment of epilepsy can be more successful after "priming" (preparing) the brain using BS as a short-term neuromodulation treatment. The limitation of testing this hypothesis is the invasive aspect of the most used classic vagal nerve stimulation (VNS) treatment for epilepsy, but the recent development of transcutaneous vagal nerve stimulation (tVNS) offered a possibility to combine chemical and electrical modulation in an earlier stage of disease, which is not tested before. The investigators want to determine the priming effect on the epileptic brain of tVNS, to make it more susceptible to add-on treatment with Brivaracetam (BRV), an AED. In addition, the investigators aim to visualize these changes in the brain because of priming, possibly altered network-organisation.

DETAILED DESCRIPTION:
Background of the study: The most prevalent neurological disorder with also immense burden of disease, epilepsy, is in over 30 percent of patients difficult to treat. The ideal treatment regime would give complete control of disease in an early stage, not only for patient well-being, but also to prevent the onset of persistent pathologic epileptic networks in the brain. The first step in treatment is the trial, and error, of multiple anti-epileptic drugs (AEDs), while invasive brain stimulation (BS) techniques with network modulating properties are saved as a last resort. The investigators hypothesize that pharmacotherapeutic treatment of epilepsy can be more successful after "priming" (preparing) the brain using BS as a short-term neuromodulation treatment. The limitation of testing this hypothesis is the invasive aspect of the most used classic vagal nerve stimulation (VNS) treatment for epilepsy, but the recent development of transcutaneous vagal nerve stimulation (tVNS) offered a possibility to combine chemical and electrical modulation in an earlier stage of disease, which is not tested before.

Objective of the study: Determine the priming effect on the epileptic brain of tVNS, to make it more susceptible to add-on treatment with Brivaracetam (BRV), an AED. In addition, the investigators aim to visualize these changes in the brain because of priming, possibly altered network-organisation.

Study design: Randomized Controlled Trial. Study population: Adults with a refractory (continuing of seizures despite 2 tried AEDs) focal epilepsy and therefore have an indication for start of Brivaracetam. Intervention (if applicable): One group receives transcutaneous vagal nerve stimulation (tVNS) 4 hours daily for the first 3 months of brivaracetam treatment. Primary study parameters/outcome of the study: Scoring on a composite index combining seizure reduction, improvement of cognition and quality of life. Secondary study parameters/outcome of the study (if applicable): Seizure reduction, seizure freedom rates, seizure severity, cognition, mood state, adverse events tVNS and brivaracetam, change in brain network properties.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable): Besides minor temporary side effects no risk is attributed to tVNS. Because of the study one extra visit is necessary, besides regular clinical follow-up. The 3 visits do require some more time than usual because of the questionnaires, MRI and short cognitive tests. The burden of the telephone calls is very limited, since it only consists of a few short questions. Patients with claustrophobia are excluded, but the requirement of lying still can be somewhat uncomfortable. The eye tracking device uses a camera in the video screen, with no burden at all.

ELIGIBILITY:
Inclusion Criteria:

* Focal epilepsy which is refractory (at least 2 different AEDs tried) and therefore has an indication for start of brivaracetam
* Age ≥ 18 years.
* IQ > 70 defined as any form of secondary education

Exclusion Criteria:

* - Inclusion not possible within 2 weeks after start of brivaracetam
* History of a progressive cerebral disorder (neurodegenerative diseases, tumours)
* History of psychogenic nonepileptic seizures (PNES)
* Inability to provide informed consent
* Any contra-indication for brivaracetam
* Current or recent use (exposed ≤ 90 days)
* Current or recent use (exposed ≤ 90 days) of levetiracetam
* Current treatment with neurostimulation
* Inability of handling the tVNS device personally
* Subjects that have a current diagnosis of cardiac arrhythmic disease
* Any contraindication for tVNS: pregnancy, active implants (such as cardiac pacemakers of cochlear implants) or cerebral shunts (e.g. ventriculo-peritoneal shunts with valve)
* Any contraindication for MRI: metallic foreign body, pacemaker, claustrophobia, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Epilepsy frequency | 6 months
  Seizure reduction (in % at 3 and 6 months in respect to baseline)
Epilepsy frequency | 6 months
  Seizure freedom rates (defined as the percentage of subjects with 100% reduction from baseline seizure frequency)
Seizure severity | 6 months
  Assessed by the National Hospital Seizure Severity Scale - NHS3, comparing scores at 3 and 6 months to baseline). Score range 1-27 (higher score = more severe).

SECONDARY OUTCOMES:
Brain networks | 3 months
  Detect changes in network properties by comparing fMRI (functional MRI) data at 3 months with baseline (independent component analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Marian M Majoie, Prof. Dr., Principal Investigator — ACE Kempenhaeghe
Locations (1):
- Stichting Kempenhaeghe, Heeze, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/16/NCT05180916/Prot_000.pdf